CLINICAL TRIAL: NCT04226690
Title: Safety of Acute and Repeated Doses of Natural Medical Marijuana Products and Effects on Subjective and Physiological Responses to Stress and Pain
Brief Title: Safety and Effects on Responses to Stress and Pain of Natural Medical Marijuana Products
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Connecticut Pharmaceutical Solutions (Unknown)
Responsible Party: Principal Investigator, RAJITA SINHA, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000020896; No NIH funding (Other: 1.19.24)
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo controlled, parallel group design
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active Dose 1 (Experimental): Participants will receive the most tolerable CBD/THC dose with repeated dosing for 7 days. On day 1 and 6/7 of the 7-day dosing, subjects will complete laboratory sessions.
  Interventions: Drug: Active CBD/THC Dose 1
- Matching Placebo (Placebo Comparator): Participants will receive a placebo with repeated dosing for 7 days. On day 1 and 6/7 of the 7-day dosing, subjects will complete laboratory sessions.
  Interventions: Drug: matched placebo comparator
- Active Dose 2 (Experimental): Participants will receive the second most tolerable CBD/THC dose with repeated dosing for 7 days. On day 1 and 6/7 of the 7-day dosing, subjects will complete laboratory sessions
  Interventions: Drug: Active CBD/THC Dose 2

INTERVENTIONS:
Drug: Active CBD/THC Dose 1 — Subjects will self-administer the assigned study medication daily at home after pickup and will be tested using medication compliance procedures. Subjects will visit the center 2 times in the 7-day period on days 1 and 7 for blood draws to assess medication compliance.
  Other Names: Medical marijuana medicine
  Arms: Active Dose 1
Drug: Active CBD/THC Dose 2 — Subjects will self-administer the assigned study medication daily at home after pickup and will be tested using medication compliance procedures. Subjects will visit the center 2 times in the 7-day period on days 1 and 7 for blood draws to assess medication compliance.
  Other Names: Medical marijuana medicine
  Arms: Active Dose 2
Drug: matched placebo comparator — Subjects will self-administer the assigned study medication daily at home after pickup and will be tested using medication compliance procedures. Subjects will visit the center 2 times in the 7-day period on days 1 and 7 for blood draws to assess medication compliance.
  Other Names: Placebo
  Arms: Matching Placebo

SUMMARY:
This proposal aims to systematically examine the safety and pharmacokinetic/pharmacodynamic profile and the physiologic, neuroendocrine and behavioral stress and pain responses to acute single doses and repeated dosing of oral tablet formulation of natural Cannabidiol (CBD) alone and in combination with Tetrahydrocannabinol and matched Placebo (PLA).

DETAILED DESCRIPTION:
This proposal aims to systematically examine the safety and pharmacokinetic/pharmacodynamic (PK/PD) profile and the physiologic, neuroendocrine and behavioral stress and pain responses to acute single doses and repeated dosing of oral tablet formulation of natural Cannabidiol (CBD) at 40 mg and 100 mg alone and in combination with Tetrahydrocannabinol (THC) at 10, 20 and 30 mg, and matched Placebo (PLA) under the following specific aims:

Aim 1: To assess the safety and PK/PD profile of acute single doses of natural oral tablet of CBD (40 mg, 100 mg), and the CBD/THC combination (40/10, 40/20 and 100/30 mg) and matching placebo (PLA) over six separate sessions one week apart in healthy adult men and women who are current recreational cannabis users (STUDY 1).

Aim 2: To examine the effects of separate CBD, THC, CBD/THC combination vs. PLA on subjective, physiological, neuroendocrine, cognitive and behavioral measures of stress, pain and anxiety at baseline and under acute pain provocation using an adapted Cold Pressor Test (CPT) in STUDY 1.

Aim 3: To examine the safety and tolerability of the two specific doses of CBD/THC, selected on the basis of best PK/PD and tolerability profile from Study 1 vs. PLA on baseline and CPT provoked pain in individuals with chronic pain over a 7-day repeated dosing (STUDY 2).

Study 1:

Eight 21-45-year-old men and women , who are recreational marijuana users but do not meet criteria for moderate-severe cannabis use disorder will be recruited to complete six separate inpatient laboratory sessions one week apart during which they will be assigned to receive an acute dose of either 40 mg CBD or 100 mg CBD alone, a CBD/THC combination of 40/10, 40/20 or 100/30 or PLA, in a random, counter-balanced, double-blind, cross-over design over a 6-week period. Sessions will be completed one -week apart to allow for an adequate washout period between sessions.

Study 2:

Adult men and women ages 21-60 (N=24) with chronic pain (not fully controlled by opioid pain medication), will be recruited and randomly assigned to receive the two most tolerable CBD/THC doses (two active doses of n=8 in each) or PLA (n=8) repeated dosing for 7 days. On day 1 and day 6/7 of the 7-day dosing, subjects will complete laboratory sessions. For 14 days after the 7-day dosing, subjects will complete daily ratings of pain and other patient-related outcomes. Subjects cannot meet criteria for moderate to severe levels of cannabis use disorder or other substance use disorders.

This registration will focus on Study 2.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and write English;
2. Recreational cannabis use with a minimum history recent use of at least one joint of smoked marijuana or marijuana edible or other equivalent form;
3. Current chronic pain, as defined by the International Classification of Diseases (ICD)-10, and stabilized for a minimum of 2 weeks on pain medication, (minimum pain ratings of 4 on a 10-point scale) and agree to not change pain medication during course of the study;
4. Body Mass Index (BMI) in the 18-36 range;

Exclusion Criteria:

1. Any psychotic disorder or current psychiatric symptoms requiring specific attention, including active symptoms of psychosis or suicidal/homicidal ideation.
2. Any Current moderate/severe Substance Use Disorder, including alcohol and cannabis.
3. Women who are nursing or have premenstrual dysphoric disorder;
4. Women who are pregnant as determined by the urine pregnancy test at each assessment period;
5. Inability to give informed consent;
6. Traumatic brain injury or loss of consciousness;
7. Individuals with current or past history of seizure disorders;

Ages: 21 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Pain Ratings | Day 1 and 7 provocation during 7-day treatment period
  Change in provoked pain ratings on day 1 and day 7 on visual analog scale of pain (range 0-10)

SECONDARY OUTCOMES:
Anxiety Ratings | Day 1 and 7 provocation during 7-day treatment period
  Change in provoked anxiety ratings on day 1 and day 7 on visual analog scale of anxiety (range 0-10)

OTHER OUTCOMES:
Pain Intensity Ratings | Baseline, 7-day treatment period and during 2 week follow-up
  Pain intensity ratings from Brief Pain Inventory (intensity range: 0-10)
Sleep disturbance Ratings | Baseline, 7-day treatment period and during 2 week follow-up
  Sleep disturbance T score from PROMIS29 sleep questions (standardized T score distribution)

CONTACTS AND LOCATIONS:
Locations (1):
- The Yale Stress Center: Yale University, New Haven, Connecticut, United States